CLINICAL TRIAL: NCT02348580
Title: Active Learning Methods for Social and Financial Education in Rwanda's Primary and Secondary Schools: A Cluster Randomized Controlled Trial
Brief Title: Effectiveness Study of Teacher Training and Social and Financial Education in Rwanda's Primary and Secondary Schools
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stichting Child Savings International (Other)
Collaborators: Association of Microfinance Institutions in Rwanda (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: TOUN-2013-Rwanda-AMIR01
Record Dates: First submitted 2014-07-09; First posted 2015-01-28 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Active Learning Methods and Life-skills Education
Keywords: teaching; education; active learning; time on task; financial education; social education; rights based education; primary school; life-skills
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment as usual (No Intervention): Schools in which regular curriculum is delivered and teachers do not receive any additional training in child centered methodologies.
- Child centered teaching of life-skills (Experimental): Training of teachers and weekly implementation of hour long sessions based on child centered teaching of life-skills education over the course of the school year in P6 and S3 classes as designed by Aflatoun Stichting Child Savings International and the Association of Microfinance Institutions in Rwanda (AMIR). The life-skills curriculum is known as Aflatoun's Child Social and Financial Education program. The training of teachers element of the intervention is known as Aflatoun Academy, which trains teachers in active learning, child centered methodologies as well as how to implement the life-skills curriculum of Aflatoun Child Social and Financial Education.
  Interventions: Behavioral: Child centered teaching of life-skills

INTERVENTIONS:
Behavioral: Child centered teaching of life-skills — The intervention includes five core components: (1) personal understanding and exploration, (2) rights and responsibilities, (3) savings and spending, (4) planning and budgeting, and (5) social and financial enterprise. The training and curriculum are both manualized. The curriculum is in English and is regionally specific (for Anglophone Africa) and has been contextualized for Rwanda. The minimum hours required by Aflatoun's fidelity guide is 20 hours which includes 10 hours of curriculum lesson and 10 hours of learning activities (savings groups, social and financial projects, club activities etc).
  Other Names: Aflatoun Child Social and Financial Education; Aflatoun Academy; Social and Financial Education; AflaAcademy; Innovation for Education
  Arms: Child centered teaching of life-skills

SUMMARY:
The study uses experimental methods to evaluate the effectiveness of an educational intervention in Rwanda. The intervention, designed by Aflatoun and AMIR, involves training teachers on the use of active-learning methods to implement a social and financial education curriculum with students in primary and secondary schools. Teachers then implement the social and financial curriculum with students in order to improve their personal, social, and financial competencies.

Teacher training will take place in November-December 2013 and the curriculum implementation will be evaluated in the 2014 school year.

The study will examine the following hypotheses:

1. Did teachers use of active learning methods in class increase due to the training received?
2. Did students' levels of engagement and on-task behaviour increase as a result of the intervention's pedagogy and content?
3. Did the following competencies of students improve due to the intervention?

   1. Self-efficacy
   2. Social skills
   3. Financial literacy
   4. Planning attitudes
   5. Savings attitudes
   6. Savings behavior
   7. Entrepreneurship
4. Did the intervention change student's pass rates on the primary six (P6) and secondary three (S3) final examinations for the classes in which it was implemented?
5. Did the intervention change student drop out rates in the classes which it was implemented?

ELIGIBILITY:
Inclusion Criteria:

* Schools willing to participate in the intervention.
* Classes of students in grade P6 or S3 during academic year 2014
* Teachers of entrepreneurship, social studies, or mathematics

Exclusion Criteria:

* Non-consenting individuals

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1750 (Actual)
Dates: Start 2013-09; Primary Completion 2014-11 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in Teacher Use of Active Learning Methods (Observed) | Up to 12 months
  A composite, standardized variable combining 5-items from an observational instrument filled out by enumerators observing teachers' classes.
Change in Teacher Use of Active Learning Methods (Self-reported) | Up to 8 months
  A composite, standardized variable combining 7-items from a self-reported instrument capturing the confidence of teachers using these seven specified active learning methods.
Change in Teacher Use of Active Learning Methods (Student report) | Up to 8 months
  A composite, standardized variable combining 4-items from students' structured interviews about their teacher's use of active learning methods.
Change in Classroom Level of Student Engagement (Observed) | Up to 12 months
  A composite, standardized variable combining structured observations of 7 randomly selected students for three different 10-second intervals in each teacher's classroom using an adapted version of the PreQuip tool designed by Educans at the University of Amsterdam.
Change in Student engagement (Student report) | Up to 8 months
  A composite, standardized variable combining 4-items measured using structured interviews of 7 randomly selected students in each teacher's classroom.

SECONDARY OUTCOMES:
Change in Students' Generalized Self-efficacy Scale (GSES-10) | Up to 8 months
  A composite, standardized variable generated based on the average sum scores of students on the GSES-10. The original four answer choice format has been changed to a five option format of (strongly disagree, disagree, neither disagree nor agree, agree and strongly agree).
Change in Students' Pro-Social (PS) (6-item) and Conduct Disorder (CD) (6-item) subscales of the Strengths and Difficulties Questionnaire (SDQ) | Up to 8 months
  A composite, standardized variable generated based on the average sum scores of students on the SDQ-CD and SDQ-PS. The original four answer choice format has been changed to a five option format of (strongly disagree, disagree, neither disagree nor agree, agree and strongly agree).
Change in Students' Financial Literacy | Up to 8 months
  A composite, standardized variable combining 4-items from student structured interviews about their financial competencies.
Change in Students' Planning Attitudes | Up to 8 months
  A composite, standardized variable combining 5-items from student structured interviews about their planning attitudes.
Change in Students' Savings Behavior | Up to 8 months
  A composite, standardized variable combining 5-items from student structured interviews about their savings behavior.
Change in Students' Savings Attitudes | Up to 8 months
  A composite, standardized variable combining 4-items from student structured interviews about their savings attitudes.
Change in Students' Entrepreneurship Attitudes & Behavior | Up to 8 months
  A composite, standardized variable combining 4-items from student structured interviews about their entrepreneurship attitudes and behavior.

OTHER OUTCOMES:
Difference in standardized examination pass rates on primary 6 (P6) and secondary 3 (S3) tests in study classes | December 2014
  Comparing the standardized test passing rates of the control and experimental group after the end of the first year of the program.
Difference in percentage drop out rates of students in study classes | December 2014
  Comparing the drop out rate of students in classes in the control and experimental group after the end of the first year of the program.
Change in Teachers use of Active Learning Methods (Observed) mediates Student Engagement (Observed) | Up to 12 months
  A mediation analysis to determine if increases in teachers use of active learning methods mediates an increase in student engagement in class.
Change in Student Engagement (Observed) mediates Students' change in Savings Behavior | Up to 12 months
  A mediation analysis to determine if increases in students' observed engagement mediates an increase in their savings behavior.

CONTACTS AND LOCATIONS:
Locations (1):
- Association of Microfinance Institutions in Rwanda, Kigali, Kigali, Rwanda